CLINICAL TRIAL: NCT00006229
Title: A Phase II/III Double Blind Randomized Trial of BMS-275291 vs. Placebo in Patients Receiving Paclitaxel/Carboplatin Chemotherapy for the Treatment of Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Paclitaxel + Carboplatin With/ut BMS-275291 in Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR18; CAN-NCIC-BR18 (Other: PDQ); BMS-CA161-003 (Other: Bristol-Myers Squibb); CDR0000068153 (Other: PDQ)
Record Dates: First submitted 2000-09-11; First posted 2003-07-25 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; N-((2S)-2-mercapto-1-oxo-4-(3,4,4- trimethyl-2,5-dioxo-1-imidazolidinyl)butyl)-L-leucyl-N,3- dimethyl-L-Valinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BMS-275291 (Experimental)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: rebimastat
- Placebo (Placebo Comparator)
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: rebimastat
  Arms: BMS-275291

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether paclitaxel and carboplatin are more effective with or without BMS-275291 for non-small cell lung cancer.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of paclitaxel and carboplatin with or without BMS-275291 in treating patients who have advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with advanced or metastatic non-small cell lung cancer treated with paclitaxel and carboplatin with or without BMS-275291.
* Compare the incidence of grade 2 or higher drug related arthritis, arthralgia and/or myalgia in patients treated with these regimens. (Phase II only)
* Compare the objective tumor response rate, time to response, and response duration in patients treated with these regimens.
* Compare the nature, severity, and frequency of toxic effects of these regimens in these patients.
* Compare the progression free survival of patients treated with these regimens. (Phase III only)
* Correlate the expression of serum/plasma and tissue matrix metalloproteinases (MMP) levels and other markers with outcomes and response in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to center, disease stage (IIIB vs IV), and ECOG performance status (0-1 vs 2). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 plus oral BMS-275291 daily on days 1-21.
* Arm II: Patients receive paclitaxel and carboplatin as in arm I plus oral placebo daily on days 1-21.

Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. BMS-275291 or placebo continues beyond 8 courses in the absence of disease progression.

Quality of life is assessed.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 776 patients will be accrued for this study within 27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIIB or IV non-small cell lung cancer (NSCLC)

  * Local or metastatic failure after surgery and/or radiotherapy allowed
* Phase II only:

  * At least one measurable lesion

    * At least 20 mm by conventional techniques OR 10 mm by spiral CT scan
* No known CNS metastases unless asymptomatic and at least 4 weeks since prior corticosteroid therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2 times ULN (5 times ULN for liver metastases)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No significant cardiac disease
* No uncontrolled high blood pressure, unstable angina, congestive heart failure, second or third degree atrioventricular conduction defects, or ventricular arrhythmias requiring medication
* No myocardial infarction within the past year

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction to drugs containing Cremophor EL
* No serious active infection or other underlying medical condition that would preclude study participation
* No peripheral neuropathy
* No condition (e.g., psychological, geographical) that would preclude study participation
* No prior breast cancer or melanoma
* No other prior malignancy within the past 5 years except carcinoma in situ, basal cell or squamous cell skin cancer, or other cancer that has been curatively treated surgically

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No prior biological response modifiers
* No other concurrent biologic therapy or immunotherapy

Chemotherapy:

* No prior antineoplastic chemotherapy, including intrapleural chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to study lesion (unless evidence of disease progression) or to 30% or greater of marrow bearing bones
* At least 1 week since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior major surgery
* No concurrent surgery

Other:

* At least 2 weeks since prior investigational drugs
* No other concurrent cytotoxic anticancer therapy
* No other investigational drugs during and for 30 days after study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2000-04-04 (Actual); Primary Completion 2003-12-10 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Smylie, MD, MB, ChB, Study Chair — Cross Cancer Institute at University of Alberta
Locations (69):
- United States (18):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Scripps Clinic, La Jolla, California
  - Central Georgia Hematology Oncology, P.C., Macon, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Carle Cancer Center, Urbana, Illinois
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Creighton University Cancer Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Erlanger Health Systems, Chattanooga, Tennessee
  - Memorial Hospital Cancer Center - Chattanooga, Chattanooga, Tennessee
  - Williamson Medical Center, Franklin, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Division of Medical Oncology - Vanderbilt, Nashville, Tennessee
- Austria (2):
  - AKH Vienna, Vienna (Wien)
  - Allgemeines Krankenhaus der Stadt Wien, Vienna (Wien)
- Belgium (3):
  - Universiteit Gent, Ghent
  - Centre Hospitalier Regional de la Citadelle, Liege (Luik)
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- Canada (17):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Helsinki University Central Hospital, Helsinki, Finland
- France (7):
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Avicenne, Bobigny
  - CHR de Grenoble - La Tronche, Grenoble
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Hopital de Neuhof, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
- Germany (5):
  - Stadisches Krankenhaus Martha Maria Halle-Dolau, Halle
  - Allgemeines Krankenhaus, Hamburg
  - Lungenklinik Hemer, Hemer
  - Marienhospital/Ruhr University Bochum, Herne
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich (Muenchen)
- Italy (5):
  - Oncologia Medica - Perugia, Perugia
  - Ospedale San Filippo Neri, Rome
  - Ospedale Carlo Forlanini, Rome
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Ospedale Civile San Giovanni e Paolo, Venezia
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Medical University of Gdansk, Gdansk, Poland
- Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia, Portugal
- Spain (3):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Servicio De Oncologia, Valencia
- Switzerland (3):
  - Kantonspital Aarau, Aarau
  - Inselspital, Bern, Bern
  - Universitaetsspital, Zurich
- United Kingdom (2):
  - Charing Cross Hospital, London, England
  - Chelsea Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradbury PA, Twumasi-Ankrah P, Ding K, et al.: The impact of brain metastases on overall survival (OS) in National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) clinical trials (CT) in advanced non-small cell lung cancer (NSCLC). [Abstract] J Clin Oncol 27 (Suppl 15): A-8075, 2009.
- [Background] Asmis TR, Ding K, Seymour L, Shepherd FA, Leighl NB, Winton TL, Whitehead M, Spaans JN, Graham BC, Goss GD; National Cancer Institute of Canada Clinical Trials Group. Age and comorbidity as independent prognostic factors in the treatment of non small-cell lung cancer: a review of National Cancer Institute of Canada Clinical Trials Group trials. J Clin Oncol. 2008 Jan 1;26(1):54-9. doi: 10.1200/JCO.2007.12.8322. PMID 18165640
- [Background] Wheatley-Price P, Le Maître A, Ding K, et al.: The influence of sex on efficacy, toxicity and delivery of treatment in National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) non-small cell lung cancer (NSCLC) chemotherapy trials. [Abstract] J Clin Oncol 26 (Suppl 15): A-8054, 2008.
- [Background] Hicks L, Cheung M, Hasan B, et al.: Venous thromboembolism and non-small cell lung cancer: a pooled analysis of National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) trials. [Abstract] Blood 110 (11): A-3995, 2007.
- [Background] Douillard JY, Peschel C, Shepherd F, Paz-Ares L, Arnold A, Davis M, Tonato M, Smylie M, Tu D, Voi M, Humphrey J, Ottaway J, Young K, Vreckem AV, Seymour L. Randomized phase II feasibility study of combining the matrix metalloproteinase inhibitor BMS-275291 with paclitaxel plus carboplatin in advanced non-small cell lung cancer. Lung Cancer. 2004 Dec;46(3):361-8. doi: 10.1016/j.lungcan.2004.05.009. PMID 15541822
- [Result] Leighl NB, Paz-Ares L, Douillard JY, Peschel C, Arnold A, Depierre A, Santoro A, Betticher DC, Gatzemeier U, Jassem J, Crawford J, Tu D, Bezjak A, Humphrey JS, Voi M, Galbraith S, Hann K, Seymour L, Shepherd FA. Randomized phase III study of matrix metalloproteinase inhibitor BMS-275291 in combination with paclitaxel and carboplatin in advanced non-small-cell lung cancer: National Cancer Institute of Canada-Clinical Trials Group Study BR.18. J Clin Oncol. 2005 Apr 20;23(12):2831-9. doi: 10.1200/JCO.2005.04.044. PMID 15837997
- [Result] Leighl NB, Shepherd F, Paz-Ares L, et al.: Randomized phase II-III study of matrix metalloproteinase inhibitor (MMPI) BMS-275291 in combination with paclitaxel (P) and carboplatin (C) in advanced non-small cell lung cancer (NSCLC): NCIC-CTG BR.18. [Abstract] J Clin Oncol 22 (Suppl 14): A-7038, 626s, 2004.